CLINICAL TRIAL: NCT01403298
Title: Project RAP: Family-based HIV Prevention in the Juvenile Drug Court
Acronym: Project RAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5K23DA021532 (NIH)
Record Dates: First submitted 2011-03-28; First posted 2011-07-27 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: HIV/AIDS
Keywords: Adolescent; HIV; AIDS; Sexual risk; Family; Prevention; Juvenile Drug Court; Juvenile Justice; Drug Use; Marijuana
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adolescent Only Health Promotion (Active Comparator): An individual adolescent-only health education program that focuses on risk behaviors related to HIV/AIDS, smoking, diet and exercise
  Interventions: Other: Adolescent Only Health Promotion
- Family-Based HIV prevention (Experimental): This individual, family-based intervention provides sex and HIV/AIDS education as part of a family-based general health education program that focuses on safe decision-making and how to control emotions to stay safe and improve parenting skills.
  Interventions: Behavioral: Family-Based HIV prevention

INTERVENTIONS:
Behavioral: Family-Based HIV prevention — This individual, family-based intervention provides sex and HIV/AIDS education as part of a family-based general health education program that focuses on safe decision-making and how to control emotions to stay safe and improve parenting skills.
  Arms: Family-Based HIV prevention
Other: Adolescent Only Health Promotion — An individual, adolescent-only health education program that focuses on risk behaviors related to HIV/AIDS, smoking, diet and exercise
  Arms: Adolescent Only Health Promotion

SUMMARY:
The purpose of this project is to compare the effect of a family-based HIV prevention program to the effect of an adolescent-only health promotion program on adolescent HIV risk and marijuana use among adolescents enrolled in the Juvenile Drug Court (JDC) of the Rhode Island Family Court.

DETAILED DESCRIPTION:
Adolescents and parents admitted to our study receive either an adolescent-only health education program that focuses on general health risk behaviors related to HIV/AIDS, smoking, diet and exercise or one that focuses on family-based HIV/AIDS education through safe decision-making and control of one's emotions as well as parent-child interactions that are associated with dysregulated affect, subsequent parenting deficits and adolescent HIV risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* 13 to 18 years old;
* male and female;
* in Rhode Island Family Court - Intake and Juvenile Drug Court program;
* English speaking

Exclusion Criteria:

* HIV infection (by self-report);
* history of sex crimes,
* current pregnancy

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
adolescent HIV/STD risk | 3 months post intervention
  Adolescent self-report of rates of condom use, number of sex partners, number of unprotected vaginal and/or anal intercourse episodes, frequency of alcohol use during sexual activity, frequency of marijuana use during sexual activity, frequency of other drug use during sexual activity
adolescent substance use | 3 months post-intervention
  Adolescent self-report of quantity and frequency of marijuana use, alcohol use and other drug use over the past 3 months and over the past 30 days. Collateral urine toxicology screen data will also be available for analysis.

SECONDARY OUTCOMES:
Scores on measures of parent-child communication (general and sex-specific),parental monitoring and family emotional environment | 3 months post intervention
  Using well-established parenting and family-based measures, such as the Parental Knowledge scales (for monitoring), Parent-Child Communication Scales (general and sexually-specific), and the Family Assessment Device (FAD), we will be obtaining both parent and adolescent report of these constructs.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Tolou-Shams, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States